CLINICAL TRIAL: NCT04207736
Title: The INVIGORATE Trial: A Randomized, Double-masked, Crossover Design, Vehicle-controlled Phase 3 Clinical Trial to Assess the Efficacy and Safety of Reproxalap Ophthalmic Solution (0.25%) Compared to Vehicle in Subjects With Seasonal Allergic Conjunctivitis Using the Environmental Exposure Chamber (EEC)
Brief Title: The INVIGORATE Trial: A Clinical Trial to Assess the Efficacy and Safety of Subjects With Seasonal Allergic Conjunctivitis.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aldeyra Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ADX-102-AC-017
Record Dates: First submitted 2019-12-19; First posted 2019-12-23 (Actual); Results first posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2022-01

CONDITIONS: Allergic Conjunctivitis
Keywords: reproxalap; INVIGORATE; ADX-102
MeSH Terms: conditions — Conjunctivitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Reproxalap Ophthalmic Solution (0.25%) (Active Comparator)
  Interventions: Drug: Reproxalap Ophthalmic Solution (0.25%)
- Vehicle Ophthalmic Solution (Placebo Comparator)
  Interventions: Drug: Vehicle Ophthalmic Solution

INTERVENTIONS:
Drug: Reproxalap Ophthalmic Solution (0.25%) — Reproxalap Ophthalmic Solution (0.25%) dosed in the Environmental Exposure Chamber.
  Arms: Reproxalap Ophthalmic Solution (0.25%)
Drug: Vehicle Ophthalmic Solution — Vehicle Ophthalmic Solution dosed in the Environmental Exposure Chamber.
  Arms: Vehicle Ophthalmic Solution

SUMMARY:
The INVIGORATE Trial: A Randomized, Double-masked, Crossover Design, Phase 3 Clinical Trial to Assess the Efficacy and Safety of Subjects With Seasonal Allergic Conjunctivitis.

DETAILED DESCRIPTION:
The INVIGORATE Trial: A Randomized, Double-masked, Crossover Design, Vehicle-controlled Phase 3 Clinical Trial to Assess the Efficacy and Safety of Reproxalap Ophthalmic Solution (0.25%) Compared to Vehicle in Subjects With Seasonal Allergic Conjunctivitis Using the Environmental Exposure Chamber (EEC).

ELIGIBILITY:
Inclusion Criteria:

* be at least 18 years of age of either gender and any race
* have at least a two-year history of moderate-to-severe ragweed-induced allergic conjunctivitis based on principal investigator's judgement
* have a positive skin prick test to ragweed pollen within the past year of screening

Exclusion Criteria:

* known contraindication or hypersensitivities to any components of the investigational product medication or components
* history of uveitis, blepharitis, dry eye syndrome, herpes simplex keratitis, or herpes zoster keratitis;
* presence of any ocular infection (bacterial, viral, or fungal) or active ocular inflammation (e.g., follicular conjunctivitis, allergic conjunctivitis) within 14 days prior to screening
* presence of any chronic ocular degenerative condition or ocular inflammation that, in the opinion of the investigator, is likely to worsen over the course of the clinical trial;
* diagnosis of moderate-to-severe pinguecula or pterygium (particularly if it results in chronic erythema), Stevens-Johnson Syndrome, ocular cicatricial pemphigoid, mucous membrane pemphigoid, significant conjunctival scarring, chemical burn, herpetic or neurotrophic keratitis, Cryopyrin Associated Periodic Syndrome (CAPS), or keratoconus
* woman of childbearing potential who is pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2019-12-05 (Actual); Primary Completion 2021-02-16 (Actual); Study Completion 2021-02-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cliantha Research, Mississauga, Ontario, Canada

REFERENCES:
- [Derived] Starr CE, Nichols KK, Lang JR, Brady TC. The Phase 3 INVIGORATE Trial of Reproxalap in Patients with Seasonal Allergic Conjunctivitis. Clin Ophthalmol. 2023 Dec 13;17:3867-3875. doi: 10.2147/OPTH.S441009. eCollection 2023. PMID 38105911

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Ninety-five subjects were randomized in a crossover design trial; efficacy was assessed in an allergy chamber.
Groups:
- Reproxalap (0.25%), Then Vehicle: Subjects first received reproxalap ophthalmic solution twice in a single day. After a washout period of approximately two weeks, subjects then received vehicle ophthalmic solution twice in a single day.
- Vehicle, Then Reproxalap (0.25%): Subjects first received vehicle ophthalmic solution twice in a single day. After a washout period of approximately two weeks, subjects then received reproxalap ophthalmic solution twice in a single day.
Period: Overall Study
Arm/Group | Reproxalap (0.25%), Then Vehicle | Vehicle, Then Reproxalap (0.25%)
Started | 48 | 47
Completed | 46 | 43
Not Completed | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Reproxalap (0.25%), Then Vehicle | Vehicle, Then Reproxalap (0.25%) | Total
Number analyzed (Participants) | 48 | 47 | 95
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.3 (13.41) | 41.9 (11.13) | 41.1 (12.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 27 | 53
  Male | 22 | 20 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 6
  Not Hispanic or Latino | 44 | 45 | 89
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 10 | 7 | 17
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 9 | 19
  White | 25 | 30 | 55
  More than one race | 3 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Subject-Reported Ocular Itching Score Assessed Over 110 to 210 Minutes in the Allergy Chamber
Description: Change from baseline comparison of reproxalap to vehicle for ocular itching on a 0 to 4 scale ( 0 = none, 4 = severe). The treatment comparison was performed using a mixed model repeated measures approach for a crossover trial with two treatment periods. The model included time point, treatment, treatment period, treatment sequence, and interaction between time point and treatment as fixed effects, and subject nested within treatment sequence as a repeated measure.
Time Frame: The efficacy assessment period was 110 to 210 minutes in the allergy chamber; baseline was pre-Dose #1 for each treatment period.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Reproxalap (0.25%): Reproxalap ophthalmic solution was dosed twice in a single day.
- Vehicle: Vehicle ophthalmic solution was dosed twice in a single day.
Arm/Group | Reproxalap (0.25%) | Vehicle
Number analyzed (Participants) | 95 | 95
score on a scale | 0.94 (0.08) | 1.38 (0.08)

2. Secondary Outcome: Conjunctival Redness Score Assessed Over 12 to 212 Minutes in the Allergy Chamber
Description: Change from baseline comparison of reproxalap to vehicle for conjunctival redness on a 0 to 4 scale ( 0 = none, 4 = extremely severe). The treatment comparison was performed using a mixed model repeated measures approach for a crossover trial with two treatment periods. The model included time point, treatment, treatment period, treatment sequence, and interaction between time point and treatment as fixed effects, and subject nested within treatment sequence as a repeated measure.
Time Frame: The efficacy assessment period was 12 to 212 minutes in the allergy chamber; baseline was pre-Dose #1 for each treatment period.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Reproxalap (0.25%) | Vehicle
Number analyzed (Participants) | 95 | 95
score on a scale | 0.51 (0.03) | 0.65 (0.03)

ADVERSE EVENTS:
Time Frame: The period of time over which adverse events were collected was approximately one day for each intervention.
Arm/Group | Reproxalap (0.25%) | Vehicle
All-Cause Mortality (participants affected / at risk) | 0/91 | 0/93
Serious Adverse Events (participants affected / at risk) | 0/91 | 0/93
Other Adverse Events (participants affected / at risk) | 69/91 | 6/93
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Reproxalap (0.25%) (N=91) | Vehicle (N=93)
General disorders and administrations site conditions (General disorders) | 68 | 6
Eye disoders (Eye disorders) | 8 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-03-24): https://cdn.clinicaltrials.gov/large-docs/36/NCT04207736/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-26): https://cdn.clinicaltrials.gov/large-docs/36/NCT04207736/SAP_001.pdf